CLINICAL TRIAL: NCT03305627
Title: Optimized Perioperative Antibiotic Prophylaxis in Radical Cystectomy
Acronym: PAPRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01480
Record Dates: First submitted 2017-09-27; First posted 2017-10-10 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Radical Cystectomy; Surgical Site Infection; Urologic Cancer; Perioperative/Postoperative Complications; Antibiotic Resistant Infection; Antibiotic Side Effect; Antibiotic-associated Diarrhea
MeSH Terms: conditions — Surgical Wound Infection; Urologic Neoplasms; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short PAP (Experimental): Perioperative antibiotic prophylaxis will be stopped after 24h
  Interventions: Other: Short PAP
- Extended PAP (Active Comparator): Perioperative antibiotic prophylaxes will be continued for 48h or more (until all indwelling urinary catheters have been removed)
  Interventions: Other: Extended PAP

INTERVENTIONS:
Other: Short PAP — Perioperative antibiotic prophylaxis for 24h
  Arms: Short PAP
Other: Extended PAP — Perioperative antibiotic prophylaxis for >48h
  Arms: Extended PAP

SUMMARY:
Cystectomy with urinary diversion (ileal conduit, orthotopic ileal bladder substitute, continent catheterizable pouch) is the best treatment option for patients with muscle-invasive bladder cancer. This intervention is one of the most challenging in urology and has a high rate of postoperative complications including around 30% of postoperative infections.

Perioperative antibiotic prophylaxis (PAP) is widely accepted as a crucial preventive measure to reduce the incidence of surgical site infections (SSI). The rationale for PAP is the reduction of the local bacterial load at the site and time of intervention, and therefore a short duration of PAP of 24 to maximal 48 hours is recommended for all clean to clean-contaminated procedures..

Evidence supporting the optimal duration of PAP for radical cystectomy with urinary diversion is lacking. Based on data extrapolated from abdominal surgery, current guidelines recommend short-term PAP (≤24h) for all clean-contaminated procedures including radical cystectomy.

However, a recent evaluation revealed a significant inter-hospital variability of PAP and showed that extended use (>48h) was common in patients undergoing radical cystectomy. Importantly, this study also demonstrated that longer duration of PAP incurred higher costs and was associated with an increased rate of C. difficile colitis. A small, prospective, non-randomized study showed equal efficacy of short-term PAP in preventing postoperative infections in patients undergoing radical cystectomy with ileum conduit compared to extended PAP. Nonetheless, larger randomized clinical trials supporting these findings are lacking.

The unwarranted extended use of antibiotics is a major concern as exposure to antibiotics is a driving force for the development of (multi-) resistant bacteria and will lead to an increasing number of difficult-to-treat infections. This has been recognized on both national and international levels and is addressed within antimicrobial stewardship frameworks.

This study will compare current practice (>48h PAP, "extended PAP") with the guideline recommended approach (24h PAP, "short term PAP") in a single-centre, prospective, randomised clinical non-inferiority trial. The primary outcome is the rate of SSI within 90 days post surgery. The aim of the study is to generate currently lacking evidence allowing for an optimised PAP strategy in a challenging surgical setting.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >18 years
* Planned radical cystectomy at the Department of Urology, Bern University Hospital

Exclusion Criteria:

* Contraindications to the classes of drugs under study, e.g. known hypersensitivity or allergy to class of drugs including alternatives described in the protocol or the investigational product,
* Women who are pregnant or breast feeding (exclusion for surgery),
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Rate of Surgical Site infections (SSI) | 90 days
  Rate of surgical site infections occurring within 90 days post surgery will be calculated for each patient.
Time to event of SSI | 90 days
  Time to event of SSI (event free survival analysis)
Rate of Urinary tract infections (UTI) | 90 days
  Rate of urinary tract infections occurring within 90 days post surgery will be calculated for each patient.
Time to event of UTI | 90 days
  Time to event of UTI (event free survival analysis)

SECONDARY OUTCOMES:
Rate and type of Antibiotic associated adverse events (AEs) | 30 days
  Rates and types of antibiotic associated AEs occurring within 30 days post surgery (direct AEs such as hypersensitivity reaction, hepatotoxicity, renal toxicity etc and indirect AEs such as line associated infections, C.difficile diarrhoea) will be assessed for each patient.
Frequency of multi-drug-resistant bacteria in urinary samples | 30 days
  The frequency of multi-drug-resistant bacteria in urine samples obtained at predefined time points during the first 30 days post surgery will be calculated for each patient
Changes in fecal flora | 30 days
  Changes in the composition of the fecal flora will be assessed in fecal samples collected at pre-specified time points
Antibiotic associated costs | 30 days
  Directly antibiotic associated costs incurred during 30days post surgery will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Thurnheer, MD, Principal Investigator — Department of Infectious Diseases, University Hospital Bern
Locations (2):
- Switzerland (2):
  - Department of Infectious Diseases, University Hospital Bern, Bern
  - Department of Urology, University Hopspital Bern, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thurnheer MC, Schurmann A, Huber M, Marschall J, Wuethrich PY, Burkhard FC. Perioperative Antibiotic Prophylaxis Duration in Patients Undergoing Cystectomy With Urinary Diversion: A Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2439382. doi: 10.1001/jamanetworkopen.2024.39382. PMID 39422911